CLINICAL TRIAL: NCT04162756
Title: A Multicenter, Open-label, Expanded Access Study of KTE-X19 for the Treatment of Subjects With Relapsed/Refractory B-Cell Malignancies
Brief Title: Study of Brexucabtagene Autoleucel (KTE-X19) for the Treatment of Individuals With Relapsed/Refractory B-Cell Malignancies
Acronym: ZUMA-18
Status: Approved for marketing | Type: Expanded Access
Sponsor: Kite, A Gilead Company (Industry)
Responsible Party: Sponsor
Organization: Gilead Sciences (Industry)
Other Study IDs: KT-US-472-0118
Record Dates: First submitted 2019-11-11; First posted 2019-11-14 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: Relapse/Refractory Mantle Cell Lymphoma
MeSH Terms: conditions — Recurrence; Lymphoma, Mantle-Cell | interventions — brexucabtagene autoleucel; fludarabine; Cyclophosphamide

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Biological: Brexucabtagene Autoleucel (KTE-X19) — A single infusion of chimeric antigen receptor (CAR)-transduced autologous T cells/kg administered intravenously.
  Other Names: Tecartus™
Drug: Fludarabine — Administered per package insert
Drug: Cyclophosphamide — Administered per package insert

SUMMARY:
The primary objectives of this study are:

Cohort 1: to provide access to brexucabtagene autoleucel (KTE-X19) for individuals with relapsed or refractory (r/r) mantle cell lymphoma (MCL) until KTE-X19 is commercially available

Cohort 2: To provide access to KTE-X19 for individuals with r/r MCL whose commercially manufactured product did not meet commercial release specification(s)

DETAILED DESCRIPTION:
This is an open-label, expanded access study of KTE-X19 for the treatment of individuals with r/r B-cell malignancies. The study will consist of 2 cohorts as indicated below:

Cohort 1 will enroll individuals prior to commercial availability of KTE-X19 for the proposed indication.

Cohort 2 will enroll individuals after KTE-X19 becomes commercially available in cases when KTE-X19 does not meet commercial release specification(s).

The participants who received an infusion of KTE-X19 will be provided the opportunity to transition to a separate long-term follow-up (LTFU) study, KT-US-982-5968.

ELIGIBILITY:
Key Inclusion Criteria:

Cohort 1:

* Pathologically confirmed mantel cell lymphoma (MCL), with documentation of either overexpression of cyclin D1 or presence of t(11;14)
* Received at least one prior regimen for MCL. Prior therapy must have included:

  * Anthracycline or bendamustine-containing chemotherapy, or
  * Anti-CD20 monoclonal antibody therapy, or
  * Treatment with Bruton's tyrosine kinase inhibitor (BTKi): ibrutinib, acalabrutinib, or a BTKi in a clinical trial for r/r MCL.
* Relapsed or refractory disease, defined by the following:

  * Disease progression after last regimen, or
  * Failure to achieve a partial response (PR) or complete response (CR) to the last regimen
* Magnetic resonance imaging (MRI) of the brain showing no evidence of central nervous system (CNS) lymphoma
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Absolute neutrophil count (ANC) ≥ 1,000/uL
* Platelet count ≥ 75,000/uL
* Absolute lymphocyte count ≥ 100/uL
* Adequate renal, hepatic, pulmonary, and cardiac function defined as the following:

  * Creatinine clearance (as estimated by Cockcroft Gault formula) ≥ 60 cc/min
  * Serum alanine aminotransferase/aspartate aminotransferase (ALT)/AST) ≤ 2.5 x upper limit of normal (ULN)
  * Total bilirubin ≤ 1.5 mg/dl, except in individuals with Gilbert's syndrome
  * Cardiac ejection fraction ≥ 50%, no evidence of pericardial effusion (except trace or physiological) as determined by an echocardiogram (ECHO), and no clinically significant electrocardiogram (ECG) findings
  * No clinically significant pleural effusion
  * Baseline oxygen saturation > 92% on room air
* Females of childbearing potential must have a negative serum or urine pregnancy test. Females who have undergone surgical sterilization or who have been post-menopausal for at least 2 years are not considered to be of childbearing potential.
* At least 1 measurable lesion. Lesions that have been previously irradiated will be considered measurable only if progression has been documented following completion of radiation therapy. If the only measurable disease is lymph node disease, at least 1 lymph node should be ≥ 2 cm.

Cohort 2:

* Individuals whose commercial manufacture of KTE-X19 did not meet commercial release specification(s)

Key Exclusion Criteria:

Cohort 1:

* Presence or suspicion of fungal, bacterial, viral, or other infection that is uncontrolled or requiring intravenous (IV) antimicrobials for management.
* History of human immunodeficiency virus (HIV) infection or acute or chronic active hepatitis B or hepatitis C infection.
* History of detectable cerebrospinal fluid (CSF) malignant cells or brain metastases or with a history of CNS lymphoma, CSF malignant cells, or brain metastases
* History of CNS disorder, such as seizure disorder, cerebrovascular ischemia/hemorrhage, dementia, cerebellar disease, cerebral edema, posterior reversible encephalopathy syndrome, or any autoimmune disease with CNS involvement

Cohort 2:

* Any medical condition that, as deemed by the treating physician, may interfere with assessment of safety or efficacy of study treatment

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Kite Study Director, Study Director — Kite, A Gilead Company
Locations (9):
- United States (9):
  - Stanford Cancer Institute, Stanford, California
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Moffitt Cancer Center, Tampa, Florida
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Cleveland Clinic, Cleveland, Ohio
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Henry-Joyce Cancer Clinic, Nashville, Tennessee
  - The University of TX MD Anderson Cancer Center, Houston, Texas